CLINICAL TRIAL: NCT04156854
Title: Pathophysiologic and Outcomes Impact of the Relation of Intravascular Volume Expansion to Neuroendocrine-Renal Function Profiles in Chronic Heart Failure - Pathway to More Individualized Therapy
Brief Title: Intravascular Volume Expansion to Neuroendocrine-Renal Function Profiles in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wayne L. Miller, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-006517
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with heart failure (Experimental): Subjects admitted to the hospital for acute decompensation of chronic systolic heart failure will have a Quantitated Blood Volume Analysis blood test done
  Interventions: Diagnostic Test: Quantitated Blood Volume Analysis

INTERVENTIONS:
Diagnostic Test: Quantitated Blood Volume Analysis — Measurement of total blood volume, composed of red blood cell mass (RBCM) and plasma volume (PV) by administering low dose iodinated I-131 labeled albumin intravenously then taking blood samples at timed increments.
  Other Names: BVA

SUMMARY:
Researchers are trying learn more about how the heart and blood volume interact in subjects with heart failure and how measuring blood volume may help them develop better ways of treating and managing heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute Decompensated Chronic Heart Failure, diagnosed clinically with volume overload by the primary Heart Failure provider or Emergency Department physician and admitted to hospital.
* New York Hear Association functional class III-IVa with stage C or D Heart Failure with Left Ventricular Ejection Fraction <50%
* Intended treatment plan with intravenous loop diuretic therapy during hospitalization
* Meeting none of the Exclusion Criteria

Exclusion Criteria:

* Age < 18 years
* Having received any investigational drug or device within 30 days prior to entry into the study.
* Clinically unstable patients (e.g. systolic blood pressure < 90 mmHg, ongoing requirement for vasopressors or mechanical circulatory support, or mechanical ventilation).
* Hospitalization within three months prior to study for hemodialysis or an ongoing requirement for hemodialysis or ultrafiltration.
* Prior organ transplantation or being on a waiting list for organ transplantation
* Presence of cardiac conditions such as clinically significant cardiac valve stenosis, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or primary arterial pulmonary hypertension (Group 1 PAH).
* History of blood pressure > 190/115 mmHg or unexplained syncope within the past 3 months.
* Symptomatic carotid artery disease, known critical carotid stenosis, or stroke within the past 3 months
* Clinically significant intrinsic renal disease (eGFR <15 ml/min/1.72m2), renal artery stenosis, or history of fibromuscular dysplasia of the renal arteries
* Baseline hemoglobin < 8.5 g/dl, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) that is five times or more the upper limit of normal or bilirubin three times or more the upper limit of normal
* History of alcohol abuse within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change in total blood volume | Baseline, 1 month, 3 month, and 6 month
  Measured in milliliters
Change in red blood cell volume | Baseline, 1 month, 3 month, and 6 month
  Measured in milliliters
Change in plasma volume | Baseline, 1 month, 3 month, and 6 month
  Measured in milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Miller, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metra M, Dei Cas L, Bristow MR. The pathophysiology of acute heart failure--it is a lot about fluid accumulation. Am Heart J. 2008 Jan;155(1):1-5. doi: 10.1016/j.ahj.2007.10.011. Epub 2007 Nov 26. No abstract available. PMID 18082481
- [Background] Cody RJ, Covit AB, Schaer GL, Laragh JH, Sealey JE, Feldschuh J. Sodium and water balance in chronic congestive heart failure. J Clin Invest. 1986 May;77(5):1441-52. doi: 10.1172/JCI112456. PMID 3517066
- [Background] Gheorghiade M, Filippatos G, De Luca L, Burnett J. Congestion in acute heart failure syndromes: an essential target of evaluation and treatment. Am J Med. 2006 Dec;119(12 Suppl 1):S3-S10. doi: 10.1016/j.amjmed.2006.09.011. PMID 17113398
- [Background] Damman K, Voors AA, Hillege HL, Navis G, Lechat P, van Veldhuisen DJ, Dargie HJ; CIBIS-2 Investigators and Committees. Congestion in chronic systolic heart failure is related to renal dysfunction and increased mortality. Eur J Heart Fail. 2010 Sep;12(9):974-82. doi: 10.1093/eurjhf/hfq118. Epub 2010 Aug 4. PMID 20685688
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Background] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385
- [Background] Miller WL, Mullan BP. Understanding the heterogeneity in volume overload and fluid distribution in decompensated heart failure is key to optimal volume management: role for blood volume quantitation. JACC Heart Fail. 2014 Jun;2(3):298-305. doi: 10.1016/j.jchf.2014.02.007. Epub 2014 Apr 30. PMID 24952698
- [Background] Anand IS, Ferrari R, Kalra GS, Wahi PL, Poole-Wilson PA, Harris PC. Edema of cardiac origin. Studies of body water and sodium, renal function, hemodynamic indexes, and plasma hormones in untreated congestive cardiac failure. Circulation. 1989 Aug;80(2):299-305. doi: 10.1161/01.cir.80.2.299. PMID 2752558
- [Background] Francis GS, Goldsmith SR, Levine TB, Olivari MT, Cohn JN. The neurohumoral axis in congestive heart failure. Ann Intern Med. 1984 Sep;101(3):370-7. doi: 10.7326/0003-4819-101-3-370. PMID 6147109
- [Background] Davila DF, Nunez TJ, Odreman R, de Davila CA. Mechanisms of neurohormonal activation in chronic congestive heart failure: pathophysiology and therapeutic implications. Int J Cardiol. 2005 Jun 8;101(3):343-6. doi: 10.1016/j.ijcard.2004.08.023. PMID 15907399
- [Background] Mentz RJ, Stevens SR, DeVore AD, Lala A, Vader JM, AbouEzzeddine OF, Khazanie P, Redfield MM, Stevenson LW, O'Connor CM, Goldsmith SR, Bart BA, Anstrom KJ, Hernandez AF, Braunwald E, Felker GM. Decongestion strategies and renin-angiotensin-aldosterone system activation in acute heart failure. JACC Heart Fail. 2015 Feb;3(2):97-107. doi: 10.1016/j.jchf.2014.09.003. Epub 2014 Oct 31. PMID 25543972
- [Background] Schrier RW. Body fluid volume regulation in health and disease: a unifying hypothesis. Ann Intern Med. 1990 Jul 15;113(2):155-9. doi: 10.7326/0003-4819-113-2-155. PMID 2193561
- [Background] Androne AS, Hryniewicz K, Hudaihed A, Mancini D, Lamanca J, Katz SD. Relation of unrecognized hypervolemia in chronic heart failure to clinical status, hemodynamics, and patient outcomes. Am J Cardiol. 2004 May 15;93(10):1254-9. doi: 10.1016/j.amjcard.2004.01.070. PMID 15135699
- [Background] Miller WL, Mullan BP. Volume Overload Profiles in Patients With Preserved and Reduced Ejection Fraction Chronic Heart Failure: Are There Differences? A Pilot Study. JACC Heart Fail. 2016 Jun;4(6):453-9. doi: 10.1016/j.jchf.2016.01.005. Epub 2016 Mar 9. PMID 26970830
- [Background] Miller WL, Mullan BP. Peripheral Venous Hemoglobin and Red Blood Cell Mass Mismatch in Volume Overload Systolic Heart Failure: Implications for Patient Management. J Cardiovasc Transl Res. 2015 Oct;8(7):404-10. doi: 10.1007/s12265-015-9650-4. Epub 2015 Sep 8. PMID 26350222
- [Background] Buglioni A, Cannone V, Cataliotti A, Sangaralingham SJ, Heublein DM, Scott CG, Bailey KR, Rodeheffer RJ, Dessi-Fulgheri P, Sarzani R, Burnett JC Jr. Circulating aldosterone and natriuretic peptides in the general community: relationship to cardiorenal and metabolic disease. Hypertension. 2015 Jan;65(1):45-53. doi: 10.1161/HYPERTENSIONAHA.114.03936. Epub 2014 Nov 3. PMID 25368032
- [Background] Gupta D, Georgiopoulou VV, Kalogeropoulos AP, Dunbar SB, Reilly CM, Sands JM, Fonarow GC, Jessup M, Gheorghiade M, Yancy C, Butler J. Dietary sodium intake in heart failure. Circulation. 2012 Jul 24;126(4):479-85. doi: 10.1161/CIRCULATIONAHA.111.062430. No abstract available. PMID 22825409
- [Background] Doukky R, Avery E, Mangla A, Collado FM, Ibrahim Z, Poulin MF, Richardson D, Powell LH. Impact of Dietary Sodium Restriction on Heart Failure Outcomes. JACC Heart Fail. 2016 Jan;4(1):24-35. doi: 10.1016/j.jchf.2015.08.007. PMID 26738949
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915
- [Background] Feldschuh J. Blood volume measurements in hypertensive disease. In: Larah JH, Brenner BM, eds. Hypertension: Pathology, Diagnosis, and Management. NY, Raven Press, 1990.
- [Background] Feldschuh J, Enson Y. Prediction of the normal blood volume. Relation of blood volume to body habitus. Circulation. 1977 Oct;56(4 Pt 1):605-12. doi: 10.1161/01.cir.56.4.605. PMID 902387
- [Background] Katz SD. Blood volume assessment in the diagnosis and treatment of chronic heart failure. Am J Med Sci. 2007 Jul;334(1):47-52. doi: 10.1097/MAJ.0b013e3180ca8c41. PMID 17630592
- [Background] Fairbanks VF, Klee GG, Wiseman GA, Hoyer JD, Tefferi A, Petitt RM, Silverstein MN. Measurement of blood volume and red cell mass: re-examination of 51Cr and 125I methods. Blood Cells Mol Dis. 1996;22(2):169-86; discussion 186a-186g. doi: 10.1006/bcmd.1996.0024. PMID 8931957
- [Background] Dworkin HJ, Premo M, Dees S. Comparison of red cell and whole blood volume as performed using both chromium-51-tagged red cells and iodine-125-tagged albumin and using I-131-tagged albumin and extrapolated red cell volume. Am J Med Sci. 2007 Jul;334(1):37-40. doi: 10.1097/MAJ.0b013e3180986276. PMID 17630590
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials